CLINICAL TRIAL: NCT06185647
Title: EPINIR-BRONCHIO : Evaluation Pragmatique de l'Impact du NIrsevimab Sur le Recours Aux uRgences Pour BRONCHIOlite Evaluation in Practice of the Impact of NIrsevimab on EmeRgency Use for BRONCHIOlitis
Brief Title: Evaluation in Practice of the Impact of NIrsevimab on EmeRgency Use for BRONCHIOlitis
Acronym: EPINIR-BRONC
Status: Completed | Type: Observational
Sponsor: Hôpital Armand Trousseau (Other)
Responsible Party: Principal Investigator, CARBAJAL, Professor, Hôpital Armand Trousseau
Other Study IDs: 20231213191724
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Bronchiolitis; Respiratory Syncytial Virus (RSV); Immunization; Infection
MeSH Terms: conditions — Bronchiolitis; Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- All infants visiting the Emergency department from october 2023 to february 2024: Extraction from medical and nursing records data on the previous administration of nirsevimab and determin whether a bronchiolitis diagnosis was given in the pediatric emergency department This information was inserted systematically in the PED records on October 31st, 2023
- All infants having the diagnosis of bronchiolitis: All patients visiting the PED for bronchiolitis. Comparison of those who received previously nirsevimab and those who did not.
  Interventions: Other: No intervention. Observational retrospective study

INTERVENTIONS:
Other: No intervention. Observational retrospective study — No intervention.
  Groups: All infants having the diagnosis of bronchiolitis

SUMMARY:
In July 2023, the Food and Drug Administration approved nirsevimab (Beyfortus®), a long-acting monoclonal antibody, for passive immunization to prevent RSV-associated lower respiratory tract infection (Bronchiolitis) among infants and young children. In Europe, The European Medicines Agency approved the use of BEYFORTUS in October 2022. In France, The Haute Autorité de Santé (HAS) approved the use of BEYFORTUS in July 2023 starting in September 2023. Beyfortus is administered as a single intramuscular injection prior to or during RSV season. This single dose may provide protection during the whole RSV season.

The safety and efficacy of Beyfortus® were supported by three clinical trials (1-3). The key measure of efficacy was the incidence of medically attended RSV lower respiratory tract infection (MA RSV LRTI ) evaluated during the 150 days after Beyfortus® administration. Beyfortus® reduced the risk of MA RSV LRTI by approximately 70% to 75% relative to placebo.

The objective of this observational study is to assess in the real-world the effectiveness of nirsevimab on the Emergency Department use for bronchiolitis as well on the effectiveness of nirsevimab to reduce hospitalization and healthcare usage in France where a national campaign to administer nirsevimab to young infants stated on September 14th, 2023.

Type of study Retrospective observational study of medical records which include systematic and prospective data on nirsevimab immunization status of patients visiting the Emergency Department.

Methodology This retrospective observational study will include two data set analysis. On one part, data from all infants presenting to the emergency department and diagnosed as having bronchiolitis will be retrieved from medical and nursing records and those who had been given nirsevimab will be compared with those who did not receive this medication prior to the ED visit. On the other part, since the investigators have included nirsevimab administration in their systematic data collection on immunization of all infants visiting our ED, the investigators will use the nirsevimab immunization status of infants diagnosed as having bronchiolitis with those do not having bronchiolitis in order to assess the effectiveness (real-world effect) of nirsevimab on the ED use and hospitalization.

DETAILED DESCRIPTION:
Bronchiolitis is a very common viral lower respiratory tract infection in infants that consists of swelling of the small airway passages in the lungs. Signs and symptoms typically begin with rhinitis and cough, which may progress to tachypnea, wheezing, rales, use of accessory muscles, and/or nasal flaring. The most common etiology of bronchiolitis is respiratory syncytial virus (RSV), with the highest incidence of infection occurring between October and March in the Northern Hemisphere. RSV can cause serious disease in infants and some children and results in a large number of emergency department and physician office visits each year. Premature infants, and those with chronic lung disease of prematurity or significant congenital heart disease, are at highest risk for severe RSV disease.

Approximately 1% to 3% of children under 12 months of age in the United States are hospitalized each year due to RSV, according to the American Academy of Pediatrics. Similar figures are found in other countries. Despite the huge burden that RSV infections represents in infants, no specific effective treatment, nor an efficacious prevention strategy had been available for term and healthy infants. The only FDA-approved product to prevent severe RSV disease among infants and young children was palivizumab, a monoclonal antibody. However, the American Academy of Pediatrics (AAP) recommends palivizumab only for children with certain underlying medical conditions (comprising <5% of all infants). In July 2023, the Food and Drug Administration approved nirsevimab (Beyfortus®), a long-acting monoclonal antibody, for passive immunization to prevent RSV-associated lower respiratory tract infection among infants and young children. Beyfortus® is indicated for the prevention of RSV lower respiratory tract disease in neonates and infants born during or entering their first RSV season, and in children up to 24 months of age who remain vulnerable to severe RSV disease through their second RSV season. In Europe, The European Medicines Agency approved the use of BEYFORTUS in October 2022. In France, The Haute Autorité de Santé (HAS) approved the use of BEYFORTUS in July 2023 starting in September 2023. Beyfortus is administered as a single intramuscular injection prior to or during RSV season. This single dose may provide protection during the whole RSV season.

The safety and efficacy of Beyfortus® were supported by three clinical trials (1-3). The key measure of efficacy was the incidence of medically attended RSV lower respiratory tract infection (MA RSV LRTI ) evaluated during the 150 days after Beyfortus® administration. One trial included 1,453 preterm infants (born at greater than or equal to 29 weeks of gestational age up to less than 35 weeks of gestation) who were born during or entering their first RSV season (1). Of the 1,453 preterm infants in the trial, 969 received a single dose of Beyfortus® and 484 received placebo. Among infants who were treated with Beyfortus®, 25 (2.6%) experienced MA RSV LRTI compared with 46 (9.5%) infants who received placebo. Beyfortus® reduced the risk of MA RSV LRTI by approximately 70% relative to placebo. A second trial included 1,490 term and late preterm infants (born at greater than or equal to 35 weeks in gestational age), 994 of whom received a single dose of Beyfortus® and 496 of whom received placebo (2). Among infants who were treated with Beyfortus®, 12 (1.2%) experienced MA RSV LRTI compared with 25 (5.0%) infants who received placebo. Beyfortus® reduced the risk of MA RSV LRTI by approximately 75% relative to placebo. In a third randomized, double-blind, controlled trial assessing the safety of nirsevimab for RSV in infants with heart or lung disease or prematurity, authors reported that the safety profile of nirsevimab was similar to that of palivizumab.

Objective The objective of this observational study is to assess in the real-world the effectiveness of nirsevimab on the Emergency Department use for bronchiolitis as well on the effectiveness of nirsevimab to reduce hospitalization and healthcare usage in France where a national campaign to administer nirsevimab to young infants stated on September 14th, 2023.

Type of study Retrospective observational study of medical records which include systematic and prospective data on nirsevimab immunization status of patients visiting the Emergency Department.

Methodology This retrospective observational study will include two data set analysis. On one part, data from all infants presenting to the emergency department and diagnosed as having bronchiolitis will be retrieved from medical and nursing records and those who had been given nirsevimab will be compared with those who did not receive this medication prior to the ED visit. On the other part, since the investigators have included nirsevimab administration in our systematic data collection on immunization of all infants visiting our ED, they will use the nirsevimab immunization status of infants diagnosed as having bronchiolitis with those do not having bronchiolitis in order to assess the effectiveness (real-world effect) of nirsevimab on the ED use and hospitalization.

The investigators included in the medical and nursing records of all patients with bronchiolitis data on the previous administration of nirsevimab on Octobre 14th, 2023. They also included on October 31st, 2023 in the medical and nursing records of all children younger than 13 months visiting the ED the nirsevimab administration whatever the reason of ED visit was.

Sample calculation The investigators used the primary objective, measurement of the real-world nirsevimab effectiveness to reduce pediatric emergency department use (PED), as a target to calculate our sample population. They computed the number of subjects needed by setting the lower boundary of the effectiveness confidence interval at 20% in infants aged 0 to 6 months. They assumed a 20% incidence of bronchiolitis in infants up to one year of age visiting the PED over the bronchiolitis season, a 50% effectiveness of Beyfortus® to reduce PED use for bronchiolitis, and a 30% rate of Beyfortus® administration in the 0-6 months population. The investigators computed the variance of the screening method estimator using the delta method. With the aforementioned hypotheses, the investigators found that a minimum of 500 infants up to one year of age will be needed. Since approximately 100 infants aged 0 to 6 months visit this PED every week during the bronchiolitis season, the investigators expect to collect the needed sample using visits from October to December.

ELIGIBILITY:
Inclusion Criteria:

* All infants aged 1 year or youger visiting the emergecy department
* All bronchiolitis visiting the emergency department during the 2023-2024 season

Exclusion Criteria:

-None

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This retrospective observational study will include two data set analysis. On one part, data from all infants presenting to the emergency department and diagnosed as having bronchiolitis will be retrieved from medical and nursing records and those who had been given nirsevimab will be compared with those who did not receive this medication prior to the ED visit. On the other part, since we have included nirsevimab administration in our systematic data collection on immunization of all infants visiting our ED, we will use the nirsevimab immunization status of infants diagnosed as having bronchiolitis with those do not having bronchiolitis in order to assess the effectiveness (real-world effect) of nirsevimab on the ED use and hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 4924 (Actual)
Dates: Start 2023-10-14 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Real-world effectiveness of nirsevimab to reduce emergency use for bronchiolitis | Bronchiolitis season: Octobre 2023-February 2024
  Determination of the nirsevimab effectiveness by using the screening method and the negative-test design
Hospital resources usage of bronchiolitis patients with and without previous administration of nirsevimab | Bronchiolitis season: Octobre 2023-February 2024
  Infants presenting bronchiolitis and having received nirsevimab will be compared to those who did not receive this medication.

SECONDARY OUTCOMES:
Age distribution of bronchiolitis patients visiting the ermergency department during the 2023-2024, 2022-2023 and 2019-2020 seasons | Bronchiolitis season: Octobre 2023-February 2024
  Compared the age distributions of two previous bronchiolitis seasons with the present season to see if the use of nirsevimab has changed this age distribution.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Armand Trousseau, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hammitt LL, Dagan R, Yuan Y, Baca Cots M, Bosheva M, Madhi SA, Muller WJ, Zar HJ, Brooks D, Grenham A, Wahlby Hamren U, Mankad VS, Ren P, Takas T, Abram ME, Leach A, Griffin MP, Villafana T; MELODY Study Group. Nirsevimab for Prevention of RSV in Healthy Late-Preterm and Term Infants. N Engl J Med. 2022 Mar 3;386(9):837-846. doi: 10.1056/NEJMoa2110275. PMID 35235726
- [Background] Griffin MP, Yuan Y, Takas T, Domachowske JB, Madhi SA, Manzoni P, Simoes EAF, Esser MT, Khan AA, Dubovsky F, Villafana T, DeVincenzo JP; Nirsevimab Study Group. Single-Dose Nirsevimab for Prevention of RSV in Preterm Infants. N Engl J Med. 2020 Jul 30;383(5):415-425. doi: 10.1056/NEJMoa1913556. PMID 32726528
- [Background] Domachowske J, Madhi SA, Simoes EAF, Atanasova V, Cabanas F, Furuno K, Garcia-Garcia ML, Grantina I, Nguyen KA, Brooks D, Chang Y, Leach A, Takas T, Yuan Y, Griffin MP, Mankad VS, Villafana T; MEDLEY Study Group. Safety of Nirsevimab for RSV in Infants with Heart or Lung Disease or Prematurity. N Engl J Med. 2022 Mar 3;386(9):892-894. doi: 10.1056/NEJMc2112186. No abstract available. PMID 35235733